CLINICAL TRIAL: NCT05723692
Title: A First-In-Human, Randomized, Double-Blind, Single and Multiple Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Subcutaneously Administered ALTB-268 in Healthy Volunteers
Brief Title: A First-In-Human SAD and MAD Study to Evaluate the Safety, Tolerability, PK and PD of SC Administered ALTB-268 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AltruBio Inc. (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ALTB-268-101
Record Dates: First submitted 2023-01-20; First posted 2023-02-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Study consists of 2 parts: Part A: a single ascending dose (SAD) and Part B: multiple ascending dose (MAD).
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALTB-268 (Experimental): Subcutaneous dose in healthy volunteers
  Interventions: Biological: ALTB-268
- Placebo (Placebo Comparator): Subcutaneous dose in healthy volunteers
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ALTB-268 — monoclonal antibody
  Arms: ALTB-268
Other: Placebo — formulation buffer
  Arms: Placebo

SUMMARY:
This study with ALTB-268 will determine the safety, tolerability, pharmacokinetics and pharmacodynamics of single and multiple ascending doses of ALTB-268 in healthy volunteers.

DETAILED DESCRIPTION:
This is a Phase I, first-in-human, randomized, double-blind, single and multiple ascending dose study to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneously administered ALTB-268 in healthy volunteers. Up to 40 and 24 healthy volunteers will be recruited in single and multiple ascending doses, respectively.

The primary objective is to assess the safety and tolerability of subcutaneously (sc) administered ALTB-268 in healthy volunteers. The secondary objective is to assess the plasma pharmacokinetics of sc administered ALTB-268 in healthy volunteers. The exploratory objectives are to assess the pharmacodynamics and evaluate immunogenicity of sc administered ALTB-268 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Written Informed Consent and willingness to comply with the study restrictions.
2. Sex: male or female volunteers.
3. Age: 18 to 55 years, inclusive, at screening.
4. Body mass index (BMI): 18.0 to 32.0 kg/m2, inclusive, at screening.
5. Weight: 50 kg to 110 kg, inclusive, at screening.
6. Healthy volunteers: Healthy status as defined by the absence of evidence of any clinically significant, in the opinion of the Investigator, active or chronic disease following a detailed medical and surgical history, a complete physical examination including vital signs, 12-lead ECG, hematology, blood chemistry, serology, and urinalysis

Exclusion Criteria:

1. Males with female partners who are pregnant, lactating, or planning to become pregnant during this study or within 90 days after dosing of study drug.
2. Use of any investigational drug or device within 30 days or five half-lives whichever is longer, of the first dose of study drug.
3. Any disease which, in the opinion of the Investigator, poses an unacceptable risk to the volunteers.
4. Clinically significant history of any drug sensitivity, drug allergy, or food allergy, as determined by the Investigator (such as anaphylaxis, hepatotoxicity, or treatment with steroids or epinephrine). Confirmatory circumstances would include treatment with epinephrine or in emergency department.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Incidence of ALTB-268 Treatment-Emergent Adverse Events | through study completion, up to day 120 of the study
  Adverse events (AEs) - severity of the AEs will be graded using the most current version of the Common Terminology Criteria for AE (CTCAE) (V5.0) 5-point scale. The relationship between AEs and the study drug will be indicated as related or not related.

SECONDARY OUTCOMES:
Pharmacokinetics of ALTB-268 AUC (PK) of sc administered ALTB-268 in healthy volunteers. | through study completion, up to day 120 of the study
  Including AUC0-t, AUC0-inf, AUC0-tau
Pharmacokinetics of ALTB-268 Cmax | through study completion, up to day 120 of the study
  Maximum plasma concentration
Pharmacokinetics of ALTB-268 tmax | through study completion, up to day 120 of the study
  Time to reach Cmax
Pharmacokinetics of ALTB-268 t1/2 | through study completion, up to day 120 of the study
  Half life
Pharmacokinetics of ALTB-268 CL/F | through study completion, up to day 120 of the study
  Apparent clearance, calculated as dose/AUC0-inf
Pharmacokinetics of ALTB-268 Rac | through study completion, up to day 120 of the study
  The ratio of accumulation of a drug after repeated administration as compared to a single dose, PART B only

OTHER OUTCOMES:
Pharmacodynamics of ALTB-268 Receptor Occupancy | through study completion, up to day 120 of the study
  Receptor Occupancy will be measured using a flow cytometry based method
Exploratory Immunophenotyping Lymphocyte subsets | through study completion, up to day 120 of the study
  Lymphocyte subsets, T,B and NK cells will be assessed using a flow cytometry based method
Pharmacodynamics - change in target engagement biomarkers | through study completion, up to day 120 of the study
  inhibition of cytokine release from ex-vivo stimulated T cells and the change of soluble (free) PSGL-1 molecule

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Dickerson, MD, Principal Investigator — ICON plc
Locations (1):
- ICON Early Development Services, Lenexa, Kansas, United States